CLINICAL TRIAL: NCT02537977
Title: CD19-directed Chimeric Antigen Receptor T Cells Therapy in Relapsed/Refractory B Cell Malignancy
Brief Title: CD19-directed CAR T Cells Therapy in Relapsed/Refractory B Cell Malignancy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Responsible Party: Principal Investigator, Aibin Liang，MD，Ph.D., Director，Department of Hematology, Shanghai Tongji Hospital, Tongji University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJ1537
Record Dates: First submitted 2015-08-26; First posted 2015-09-02 (Estimated); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Leukemia; Lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CAR-T cells (Experimental): Autologous 2nd generation CD19-directed CAR-T cells
  Interventions: Biological: CD19-directed CAR-T cells

INTERVENTIONS:
Biological: CD19-directed CAR-T cells — CD19-directed CAR-T cell infusion will be given by vein

SUMMARY:
Relapsed/refractory leukemia and lymphoma lack effective treatment. The cancer immunotherapy with chimeric antigen receptor (CAR) T cells provides a potent new approach for them. In this clinical trial, the investigators aim to assess the safety and efficacy of administering T cell expressing an anti-CD19 CARs to patients with chemotherapy resistant or refractory CD19 positive B cell malignancy including leukemia and lymphoma.

DETAILED DESCRIPTION:
Tongji Hospital of Tongji University has developed an investigational approach for treating patients with CD19 positive B cell malignancy that involves taking white blood cells from the patient, growing them in the laboratory in large numbers, genetically modifying these specific cells with lentivirus to attack CD19 positive cells, and then giving the cells back to the patients.The main purpose of the study is to assess the safety and efficacy of the treatment with anti-CD19 CAR-T cells in the patients with chemotherapy resistant or refractory CD19 positive B cell malignancy including leukemia and lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CD19+ leukemia or lymphoma, meeting the following criteria:

  * At least 2 prior combination chemotherapy regimens (not including single agent monoclonal antibody (Rituximab) therapy)
  * Less than 1 year between last chemotherapy and progression
  * Not eligible or appropriate for allo-HSCT
* To be aged 6 to 85 years
* Estimated survival of ≥ 6 months, but ≤ 2 years
* ECOG score ≤2
* Relapse after auto-HSCT
* Women of childbearing potential must have a urine pregnancy test taken and proven negative prior to the treatment. All patients agree to use reliable methods of contraception during the trial period and until follow-up for the last time
* Voluntary participation in the clinical trials and sign the informed consent

Exclusion Criteria:

* History of epilepsy or other CNS disease
* Patients have GVHD, which needs treatment with immunosuppressive agents
* Patients with prolonged QT interval or severe heart disease
* Patients in pregnancy or breast-feeding period
* Uncontrolled active infection
* Active hepatitis B or hepatitis C infection
* Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary
* Previously treatment with any gene therapy products
* Feasibility assessment during screening demonstrates <20% transduction of target lymphocytes, or insufficient expansion (<5-fold) in response to CD3/CD28 costimulation
* ALT /AST>3 x normal value; Creatinine> 2.5 mg/dl; Bilirubin >2.0 mg/dl
* Any uncontrolled medical disorders that the researchers consider are not eligible to participate the clinical trial
* HIV infection
* Any situation that would increase dangerousness of subjects or disturb the outcome of the clinical study according to the researcher's evaluation

Ages: 6 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Occurrence of study related adverse events | 2 years
  defined as >= Grade 3 signs/symptoms, laboratory toxicities, and clinical events) that are possibly，likely，or definitely related to the study.

SECONDARY OUTCOMES:
Response rates to CAR-T cells | 2 years
  Describe the response rates of patients treated with CAR-T cells, including complete remission, partial remission,stable disease and progression disease
Progression free survival(PFS) | 2 years
Duration of remission(DOR) | 2 years
Overall survival(OS) of patients treated with CAR-T cells | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Aibin Liang, MD,Ph.D., Principal Investigator — Shanghai Tongji Hospital, Tongji University School of Medicine
Locations (1):
- Shanghai Tongji Hospital, Tongji University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No